CLINICAL TRIAL: NCT04170673
Title: Development of a Global Scale Assessing Impairment in Cerebral Small Vessel Diseases
Acronym: SMACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190597
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2019-11

CONDITIONS: Small Vessel Cerebrovascular Disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In daily practice, several scales are used to evaluate patients with small vessel diseases of the brain (SVD). However, these scales exclude key symptoms such as apathy and mood disorders observed in SVD. Furthermore, the use of a combination of scales does not allow neither a very sensitive assessment of clinical changes, neither an overall assessment of a patient's outcome.

Moreover, there is no scale dedicated to cognitive, emotional and behavioural complaints in patients with SVD. These patients are evaluated with scales used in neurodegenerative diseases such as Alzheimer's disease and frontotemporal dementia. These are scales that have been developed in the elderly and they are not sensitive to minor complaints. It is needful to develop scales adapted to patients with SVD in order to understand the consequences of the disease symptoms on their daily life at inclusion and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* French mother language
* French reading and writing
* The patient can fulfil the questionnaire on his own, without any help.
* Brain imaging suggestive of SVD: confluent white matter hypersignals with symmetric distribution, small deep infarction, cerebral haemorrhage, microbleeds

Optional:

• Presence of informative companion in contact with the patient at least once every 15 days

Exclusion Criteria:

* Presence of unacquired cognitive impairment (mental retardation, developmental disorders)
* Presence of non-vascular leukoencephalopathy
* Clinical picture and evolution suggesting a degenerative disease
* Serious or unstable psychiatric problems (psychoses, severe depression)
* Unstable clinical status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with small vessel disease will be recruited from the Department of Neurology at Lariboisière Hospital. The study will be proposed to patients when they come to Lariboisière Hospital for hospitalization (full hospitalization or day hospitalization) or consultation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Develop a Global Clinical Severity Scale in Patients with cerebral SVD | 3 years post-inclusion
  The primary outcome is to develop this scale, thus precise definition of the scale is not available

SECONDARY OUTCOMES:
Internal validity of each scale | 3 years post-inclusion
  To analyze correlations between items, scale structure, o floor and ceiling effects and profiles of missing data
Intra evaluator reliability | 3 years post-inclusion
Inter-evaluator reliability | 3 years post-inclusion
Scale validity | 3 years post-inclusion
Scale sensitivity to change | 3 years post-inclusion
  To determine clinically important minimal difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Lariboisiere hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided